CLINICAL TRIAL: NCT01184027
Title: Impact of Nutrition and Swallowing Function in a Randomized Controlled Trial of Head and Neck Cancer Patients During the Course of Treatment
Brief Title: Impact of Nutrition and Swallowing Function of Head and Neck Cancer Patients During the Course of Treatment
Status: Withdrawn | Type: Observational
Why Stopped: The study did not receive funding.
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Catherine Kubrak, Principal Investigator, University of Alberta
Other Study IDs: HN 11226
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Head and Neck Cancer; Surgery; Nutrition; Swallowing
Keywords: head and neck cancer; surgery; nutrition
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- G-tube/swallowing intervention: patients will receive G-tube/nutritional and swallowing intervention. As per patient needs
  Interventions: Behavioral: G-tube/swallowing intervention
- G-tube/swallowing counseling: G-tube/ad lib dietary and swallowing counseling. Current standard of care.
- nutrition/swallowing intervention: Patients will receive active nutrition and swallowing intervention based on patients caloric and swallowing needs.
  Interventions: Behavioral: nutrition /swallowing intervention
- nutrition/swallowing counseling: Patients will have ad lib dietary intake with general nutrition and swallowing counseling.
  Interventions: Behavioral: nutrition /swallowing counseling

INTERVENTIONS:
Behavioral: nutrition /swallowing counseling — general nutrition and swalling information
  Other Names: Group 4
  Groups: nutrition/swallowing counseling
Behavioral: G-tube/swallowing intervention — Patient will have active swallowing intervention with an SLP
  Other Names: Group 1
  Groups: G-tube/swallowing intervention
Behavioral: nutrition /swallowing intervention — Patient will have active (daily) nutrition and swallowing intervention based on patients individual needs.
  Other Names: Group 3
  Groups: nutrition/swallowing intervention

SUMMARY:
Weight loss resulting from poor food intake is common in head and neck cancer patients. Currently, feeding tubes are placed before starting treatment to provide nutrition and prevent weight loss. However, studies have not always shown that feeding tubes prevent weight loss. Also, limiting food intake by mouth may lead to swallowing problems. The aim of this study is to compare the effect of diet and swallowing therapy with feeding tube placement. In this study, your weight, food intake, swallowing ability, and side-effects of treatment will be monitored before, during, and 3 and 6 months after treatment to see if there is any difference between the therapy groups. The investigators hope that with the addition of diet and swallowing therapy during treatment that we can improve food intake and swallowing ability while still maintaining weight.

DETAILED DESCRIPTION:
Background: Multimodal treatment for advanced head and neck cancer (HNC) is associated with acute toxicities including mucositis, xerostomia, and dysphagia and a high prevalence of weight loss, requiring nutritional intervention. Currently, there is ongoing debate about the best way to provide nutrition support while undergoing chemoradiation (CRT) therapy after surgery for advanced head and neck cancer (HNC). Randomized controlled trials comparing the nutritional benefits of feeding tubes over dietary counseling and/or supplementation have not conclusively demonstrated a reduction in weight loss, unplanned hospitalizations, treatment toxicities, or tumour control. Additionally, the relative benefits of feeding tubes are controversial. Studies evaluating the efficacy of feeding tubes report that patients with feeding tubes have increased risk of aspiration, feeding tube dependence, a small but finite risk of tumour seeding, but more importantly long term functional swallowing impairment. However, emerging data are reporting that swallowing exercise programs that are designed to strengthen musculature throughout the course of treatment may lead to improved return of functional swallowing. Thus, preservation of functional swallowing may potentially improve return to oral nutrition.

Purpose: Our purpose of this study is to compare the efficacy of nutritional and swallowing intervention with/out a percutaneous endoscopic gastrostomy (PEG) tube to that of ad lib nutrition and swallowing counseling with/out a PEG tube in advanced HNC patients. Weight, caloric intake, instrumental swallowing function, xerostomia, mucositis, pain, unplanned treatment interruptions, unplanned hospital admissions, complications, duration of feeding tube, tumour control, performance status, and quality of life (QOL) will be assessed before, during, 3 and 6 months after CRT therapy to determine if there is any differences between the intervention groups.

Study Design: A randomized controlled longitudinal design during the entire course of treatment including surgery and CRT therapy will be conducted to investigate the efficacy of nutritional and swallowing interventions in HNC patients at baseline, after each course of consecutive course treatment and 3 and 6 month follow-up. Patients demonstrating a safe functional swallow following surgery will be randomly assigned to one of four groups: Group 1 - patients will receive PEG tube/in-depth nutrition and swallowing intervention; Group 2 - patients will receive PEG tube/ad lib nutrition and swallowing counseling; Group 3 - patients will receive in-depth nutrition and swallowing intervention; or Group 4 - patients will receive ad lib nutrition/Kaofeed tube nutrition and swallowing counseling.

Study Sample: Patients with diagnosis of HNC to the oral cavity, pharynx, and larynx undergoing surgery and CRT therapy at the University of Alberta Hospital (UAH) and Cross Cancer Institute (CCI) will be eligible for participation in the study.

Inclusion criteria are: ≥ 18 years of age; diagnosed with HNC to sites of the oral cavity, oropharynx, and larynx; all histologic types of cancer; advanced tumour stages; all forms of radiation therapy (RT) including standard or investigational for HNC; all forms of chemotherapy (CT) including standard or investigational for HNC; alert and mentally competent; English-speaking. Exclusion criteria are: unable to have safe swallow following surgical intervention; allergy or intolerance to any enteral nutritional supplements in current use; renal insufficiency. There are approximately 3-4 HNC patients scheduled for surgery, and CRT therapy per week at UAH/CCI. With a significance level of 0.01 between groups and a power of 0.85 (an effect size of 0.9) a minimum sample size of 41 patients is required for this study. As a pilot study with 20 degrees of freedom, an adequate and reasonable sample size would require 24 patients to be recruited to participate.

Data Collection: Patients will be informed of the study and consent obtained. Demographic and clinical data will be collected at the time of recruitment. Patient's height and weight will be recorded. Patients will be asked to complete the Patient Generated Subjective Global Assessment, Head and Neck Symptom Checklist, Edmonton Symptom Assessment Score and University of Washington Quality of Life Revised Questionnaire. Patients will be given instructions on how to complete the 24h dietary recall, will have assessments for mucositis and xerostomia and an appointment for modified barium swallow. After surgery, patient's who have a verified safe swallow by a speech-language pathologist (SLP) and MBS will be randomized into 1 of 4 groups. Patient randomized to Group 1 or 2 will have percutaneous gastrostomy (PEG) tubes inserted as per gastroenterology PEG tube insertion protocol. Patients randomized to Group 1 or 3 will have additional nutrition and swallowing intervention. Patients randomized to Group 3 or 4 who have symptoms that prevent them from swallowing or have a >5% weight loss during treatment will be offered a Kaofeed tube for nutrition supplementation. Nutritional intervention as outlined in studies by Ravasco et al. (2005) and Goncalves Dias et al (2005) will include individualized nutrition orientation to therapeutic diet that will aid the patient in achieving a caloric and protein intake which promotes approximately 40 kcal/kg/day. The nurse practitioner together with the patient will meet on a daily basis to review their therapeutic diet and resolve issues of symptom management that prevent dietary intake. Swallowing intervention will include evaluation of functional swallowing by a SLP. The SLP together with the patient will meet on a daily basis to review functional swallowing and will teach/aid the patient to adjust their swallowing to meet their changing safe swallowing needs. All parameters and study measurement are outlined in Table 1.

Data Analysis: Descriptive statistics will be used to generate a profile of the nutrition status, caloric intake, nutrition impact symptoms, swallowing function, quality of life, unplanned treatment interruptions, unplanned hospital admissions, and complications of HNC patients at baseline, after each course of consecutive course treatment and 3 month follow-up. Changes, as well as differences in nutrition status, caloric intake, nutrition impact symptoms, quality of life and swallowing function before and after each course of treatment, and 3 month follow-up will be examined using t-tests and analysis of variance (ANOVA).

Significance of the Study: The high prevalence and negative consequences of weight loss, primarily stemming from dysphagia in advanced HNC patients using the current multimodal treatment regime supports the need to determine the most effective nutritional management of this patient group. Additionally, this pilot study may establish the foundation for future protocols and guidelines for nutritional care of HNC patients.

ELIGIBILITY:
* Inclusion criteria are:

  * ≥ 18 years of age;
  * diagnosed with HN cancer to sites of the oral cavity, pharynx, and larynx;
  * all histologic types of cancer;
  * advanced tumour stages;
  * all forms of RT including standard or investigational for HNC;
  * all forms of CT including standard or investigational for HNC;
  * alert and mentally competent;
  * English-speaking.

Exclusion criteria are:

* unable to have safe swallow following surgery;
* allergy or intolerance to any enteral nutritional supplements in current use;
* renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Head and Neck Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
nutrition status | 6 months
  evaluation of caloric intake

SECONDARY OUTCOMES:
swallowing function | 6 months
  maintenance of swallowing function

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Kubrak, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital (Otolaryngology), Edmonton, Alberta, Canada